CLINICAL TRIAL: NCT05820672
Title: A US Multi-center, Prospective, Non-interventional, Long Term, Effectiveness and Safety Study of Patients Treated With SKYTROFA (Lonapegsomatropin)
Brief Title: A US Non-interventional, Effectiveness and Safety Study of Patients Treated With SKYTROFA
Acronym: SkybriGHt
Status: Recruiting | Type: Observational
Sponsor: Ascendis Pharma Endocrinology Division A/S (Industry)
Responsible Party: Sponsor
Organization: Ascendis Pharma A/S (Industry)
Other Study IDs: ASND0037
Record Dates: First submitted 2023-03-07; First posted 2023-04-20 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Growth Hormone Deficiency
Keywords: Human Growth Hormone; SKYTROFA
MeSH Terms: conditions — Dwarfism, Pituitary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients on SKYTROFA Treatment: Patients on SKYTROFA Treatment managed in USA with appropriate written Informed Consent
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The goal of this study is to genrate evidence on long-term effectiveness and safety of SKYTROFA (lonapegsomatropin) in patients with growth hormone deficiency under routine clinical care

DETAILED DESCRIPTION:
Patients will be treated according to routine clinical practice, and no additional visits, examinations or tests will be required beyond those performed as part of routine clinical practice except for COAs.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are on treatment with SKYTROFA (lonapegsomatropin)
* Patients being clinically managed in USA
* Patients with an appropriate written informed consent/assent as applicable for the age of the patient

Exclusion Criteria:

* Patients participating in any interventional clinical study

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients being treated with SKYTROFA who are associated to selected endocrinology or pediatric clinics across USA.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2033-03 (Estimated); Study Completion 2033-03 (Estimated)

PRIMARY OUTCOMES:
Assess the safety of patients treated with SKYTROFA (Lonapegsomatropin) | 5 years
  Incidence of Adverse Events and Serious Adverse Events
Assess the effectiveness of patients treated with SKYTROFA (Lonapegsomatropin) | 5 years
  Near adult height (cm)

SECONDARY OUTCOMES:
Assess clinical outcome assessments (COAs) | 5 years
  Change in Quality of Life in Short Stature Youth (QoLISSY) scores from baseline through End of Study (QOLISSY scores range on a scale of 0 to 100 with higher scores representing better quality of life. (For both child and parent version))
Assess clinical outcome assessments (COAs) | 5 years
  Change in Treatment Satisfaction Questionnaire for Medicine (TSQM-9) scores from baseline through End of Study (The TSQM-9 domain scores range from 0 to 100 with higher scores representing higher satisfaction on that domain)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — Ascendis Pharma A/S
Locations (26):
- United States (26):
  - Ascendis Investigational Site, Phoenix, Arizona
  - Ascendis Investigational Site, Orange, California
  - Ascendis Investigational Site, Sacramento, California
  - Ascendis Investigational Site, San Francisco, California
  - Ascendis Pharma Investigational Site, Centennial, Colorado
  - Ascendis Investigational Site, Washington D.C., District of Columbia
  - Ascendis Investigational Site, Orlando, Florida
  - Ascendis Investigational Site, Tampa, Florida
  - Ascendis Investigational Site, Sandy Springs, Georgia
  - Ascendis Investigational Site, Boise, Idaho
  - Ascendis Investigational Site, Indianapolis, Indiana
  - Ascendis Investigational Site, Iowa City, Iowa
  - Ascendis Investigational Site, Louisville, Kentucky
  - Ascendis Investigational Site, Minneapolis, Minnesota
  - Ascendis Investigational Site, Las Vegas, Nevada
  - Ascendis Investigational Site, Lebanon, New Hampshire
  - Ascendis Investigational Site, Manchester, New Hampshire
  - Ascendis Investigational Site, Morristown, New Jersey
  - Ascendis Investigational Site, New Hyde Park, New York
  - Ascendis Investigational Site, Cincinnati, Ohio
  - Ascendis Investigational Site, Portland, Oregon
  - Ascendis Investigational Site, Columbia, South Carolina
  - Ascendis Investigational Site, Dallas, Texas
  - Ascendis Investigational Site, El Paso, Texas
  - Ascendis Investigational Site, Norfolk, Virginia
  - Ascendis Investigational Site, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No